CLINICAL TRIAL: NCT03978936
Title: Improving Medication Adherence With Telehealthcare Medication Therapy Management to Change Health Outcomes in Adolescents and Young Adults With Asthma
Brief Title: Medication Adherence With Telehealthcare Medication Therapy Management
Acronym: MATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Nemours Children's Health System (Other); American Lung Association (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00197194; 1R01HL136945-01A1 (NIH); 3R01HL136945-01A1S1 (NIH)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Uncontrolled Asthma; Young Adults
Keywords: Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Obstructive Lung Diseases
MeSH Terms: conditions — Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — Medication Therapy Management; myotubularin

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, superiority trial with two intervention groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTM-EAM (Experimental): Medication Therapy Management Video Telehealthcare plus Electronic Adherence Self-Management [MTM-EAM]
  Interventions: Behavioral: Medication Therapy Management (MTM) Video Telehealthcare; Behavioral: Electronic Adherence Self-Management (EAM)
- EAM only (Active Comparator): Electronic Adherence Self-Management [EAM] only
  Interventions: Behavioral: Electronic Adherence Self-Management (EAM)

INTERVENTIONS:
Behavioral: Medication Therapy Management (MTM) Video Telehealthcare — MTM is an individualized approach to "optimize medication use for improved patient outcomes" and is designed to "empower patients to take an active role in managing patients' medications" thus, providing a favorable strategy for addressing adherence issues. Five core elements define MTM: complete medication therapy review (CMR), creation of a personal medication list (PML), development of a medication action plan (MAP), intervention and/or referral for drug therapy problems, and documentation and follow-up
  Arms: MTM-EAM
Behavioral: Electronic Adherence Self-Management (EAM) — Participants will have a sensor which monitors their adherence to medication use

SUMMARY:
Improving Medication Adherence with Telehealthcare Medication Therapy Management to Change Health Outcomes in Adolescents and Young Adults with Asthma (MATCH) is a multi-center, randomized parallel group study targeted to an at-risk population of Adolescents and Young Adults (AYA) with uncontrolled asthma who have poor adherence with prescribed Inhaled corticosteroid (ICS) therapy.

DETAILED DESCRIPTION:
The study evaluates a Medication Therapy Management (MTM) video telehealthcare intervention to address poor medication adherence. In addition, it employs a novel method to track and provide feedback to participants on adherence by using Propeller Sensors. 300 adolescents and young adults will be randomized to Medication Therapy Management (MTM) video telehealthcare plus electronic adherence self-management [MTM EAM] or electronic adherence self-management alone (EAM). Due to the hierarchal design of the trial, two primary outcomes to be tested in a sequential manner are specified, adherence and time to first asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 through 35 years
* Speaks English or Spanish
* Physician diagnosed asthma (without any other co-morbid pulmonary disease)
* Prescribed ICS treatment for at least 3 months prior to screening
* Adherence to Refills and Medication Scale (ARMS) 7-item questionnaire score of >8 (low or moderate adherence)
* Current use of albuterol metered dose inhaler (MDI) for rescue: ProAir, Ventolin, albuterol sulfate (from Prasco or Teva)
* Uncontrolled asthma:
* Symptomatic asthma defined as 3 of the following in the past 4 weeks:
* Daytime symptoms of asthma more than twice per week
* Any night awakening due to asthma
* Rescue inhaler use for symptoms more than twice per week
* Any activity limitation due to asthma; OR
* Asthma Control Test score ≤19
* Has iPhone or Android smart phone with Short Message Service (SMS)
* Has access to reliable WiFi service and a device with capability for telemedicine study visits
* Ability to understand and willingness to sign consent documents
* Evidence of Propeller sensor connection in the 4-week run-in period

Exclusion Criteria:

* Use of an investigational treatment in the previous 30 days.
* Previous enrollment in MATCH Structured Interviews ( Aim 1)
* Currently enrolled in an intervention trial
* Currently uses an ICS not compatible with the Propeller sensor
* Inability to comply with study procedures, including:
* Inability or unwillingness to provide informed consent (or assent in the case of a minor).
* Inability to perform study measurements.
* inability to be contacted by phone via calls and /or text messaging
* Not willing to have video chat
* Any condition(s) in the opinion of the physician that puts the participant at risk from participating in the study

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 321 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Time (days) to first exacerbation event | 12 months
  Time to first asthma exacerbation is the time to first exacerbation event defined as a worsening of asthma requiring the use of systemic corticosteroids for at least 3 days, or asthma-specific emergency department visit with treatment with systemic corticosteroids, or asthma-specific hospitalization, or death (all cause and asthma exacerbation). 104. These data will be collected by self-report in the "My Asthma" bi-weekly assessment questionnaire, and verified by the study site coordinator with the participant's provider.
Proportion of adherent days as assessed by Propeller sensors | 12 months
  Adherence will be measured using data collected from Propeller sensors. Adherence for each day is calculated as the number of inhalations taken divided by the expected number of doses. A day will be defined as adherent if the participant completes 80% or more of the prescribed inhalations. The primary outcome will be the proportion of adherent days over the course of follow-up, i.e. from the randomization visit to the 1-year visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Blake, Pharm.D, Principal Investigator — Nemours Children's Specialty Care; Robert Wise, MD, Principal Investigator — Johns Hopkins School of Medicine; Janet Holbrook, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (21):
- United States (21):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of California at San Francisco, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Hospitals, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - New York University School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mount Sinai National Jewish Health Respiratory Institute; Icahn School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Vermont Lung Center at The University of Vermont, Colchester, Vermont
  - Pacific Northwest Airways - VA Puget Sound Healthcare System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blake KV. Telemedicine and adherence monitoring in children with asthma. Curr Opin Pulm Med. 2021 Jan;27(1):37-44. doi: 10.1097/MCP.0000000000000739. PMID 33105234